CLINICAL TRIAL: NCT03342105
Title: The Efficacy and Safety of Cettum for Perennial Allergic Rhinitis: a Randomized, Open-label, Assessment-blind, Parallel Designed Pilot Clinical Study
Brief Title: The Efficacy and Safety of Cettum for Perennial Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eun Jung Kim (Other)
Collaborators: DongGuk University (Other)
Responsible Party: Sponsor-Investigator, Eun Jung Kim, Investigator, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUIH 2017-0013
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Rhinitis, Allergic
Keywords: Rhinitis, Allergic; Moxibustion
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cettum (Electrical moxibustion) (Experimental): The patients in this group will receive Cettum (Electrical moxibustion) treatment applied by a certified Korean Medicine Doctor with more than 6 years of traditional Korean medicine college education.
  Interventions: Procedure: Cettum
- Acupuncture (Active Comparator): The patients in this group will receive acupuncture treatment applied by a certified Korean Medicine Doctor with more than 6 years of traditional Korean medicine college education.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Cettum — The treatment will be applied in 8 sessions, 2 times per week for 4 weeks. Moxibustion will be provided at 11 standard acupuncture points: EX-HN3, and both EX-HN8, LI20, LI4, GB2, ST36. A specifically designed device, Cettum (20X28X18mm) manufactured by K-medical Co.(Korea), will be used to treat patients in this group. The expected total time of each treatment session will be 15 min.
  Other Names: Electrical moxibustion
  Arms: Cettum (Electrical moxibustion)
Procedure: Acupuncture — The treatment will be applied in 8 sessions, 2 times per week for 4 weeks. Acupuncture will be provided at same points in the Cettum group. Sterile stainless steel disposable acupuncture needles (0.25X30mm, DongBang Acupuncture Inc, Korea) will be used to treat patients in this group. The needles will be kept in place for 15 min.
  Arms: Acupuncture

SUMMARY:
The purpose of this study is verify the efficacy and safety of Cettum (Electrical moxibustion) for patients with perennial allergic rhinitis.

DETAILED DESCRIPTION:
The investigators target the patients with perennial allergic rhinitis. After treatment in 2 groups (Cettum treatment and acupuncture treatment) the investigators will compare the effects of relieving symptoms and improving quality of life. So the investigators will confirm the efficacy of Cettum, and further the best treatment method. In addition, the investigators are going to evaluate the safety of abnormal reaction during the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 60 years-old
2. Presence of nasal symptoms more than 2 consecutive years
3. Presence of two or more nasal symptoms (rhinorrhea, nasal congestion, nasal itching, and sneezing) with severity score ≥ 2 (0 = no symptoms, 1 = mild symptom(s), 2 = moderate symptom(s), and 3 = severe symptom(s))
4. Positive reaction to the one or more perennial allergen in skin prick test
5. Not having a problem with expression of opinion
6. Willingness to participate in this trial and to sign the informed consent agreement

Exclusion Criteria:

1. Treatment with nasal/oral corticosteroids within the past month; herbal medication for rhinitis within the past month; nasal cromolyn or tricyclic antidepressants within the past two weeks; nasal/oral decongestants, nasal/oral antihistamines, or antileukotrienes within the past week
2. Presence of rhinosinusitis (paranasal sinus X-ray demonstrating mucosal thickening or opacification of the paranasal sinuses)
3. Presence of neoplasm, severe systemic inflammation, or other systemic disease that affects rhinitis
4. History of anaphylaxis for allergic tests
5. Females who is pregnant or lactating
6. Being difficult to maintain treatment (e.g. paralysis, severe physical or psychiatric disorder, dementia, drug intoxication, severe visual or hearing impairment)
7. Being afraid of moxibustion treatment or expected adverse effects
8. When the investigators determine that it is inappropriate for participation

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 4 weeks
  TNSS evaluates symptoms of rhinorrhea, nasal congestion, nasal itching and sneezing on a 4-point scale. The total score range is from 0 to 12, where 0 = no symptoms, 1 = mild symptom(s), 2 = moderate symptom (s), and 3 = severe symptom(s). TNSS baseline value will be measured prior to the start of the experiment and then again during every visit.

SECONDARY OUTCOMES:
Rhinoconjunctivits Quality of Life Questionnaire (RQLQ) | 4 weeks
  RQLQ is self-report questionnaire used to assess the quality of life in patients with allergic rhinitis. The questionnaire has 7 domains; activity limitations, sleep disturbances, non-hay fever symptoms, practical problems, nasal symptoms, ocular symptoms and emotional problems. Patients will be asked to recall their experiences during the previous week and to rate each question on a ranging from 0 (no impairment) to 6 (severe impairment). RQLQ will be measured during visits 2, 6, 9, and 10.
Total serum IgE and eosinophil count levels | 4 weeks
  Total serum IgE and eosinophil count levels will be measured during visits 2 and 9.
Pre KiFDA AR version 2.0 | 4 weeks
  The investigator, traditional Korean medicine doctor, will evaluate the nasal endoscopy index during visits 2 and 9. The investigator will check the score following observation of the nasal membrane color, rhinorrhea, and inferior turbinate swelling of the patient via nasal endoscopy.
Pre KiFDA AR version 3.0 | 4 weeks
  The investigator, traditional Korean medicine doctor, will select a pattern for each patient from among lung-heat, lung-cold and spleen-qi-deficiency through face-to-face diagnoses, based on body and nasal conditions.
Adverse Events | 4 weeks
  Any unpredicted symptoms are checked at every visit and if any, the symptom, time of occurrence, and length of duration are recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Ug Hong, Ph. D., Principal Investigator — DongGuk University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jo HR, Sung WS, Jung CY, Lim CY, Lee SD, Hong SU, Kim KH, Kim EJ. Effectiveness and safety of electric heating moxibustion for perennial allergic rhinitis: A pilot, randomized, assessor-blind trial. Complement Ther Med. 2022 Sep;68:102835. doi: 10.1016/j.ctim.2022.102835. Epub 2022 Apr 22. PMID 35470006
- [Derived] Jung CY, Cho MJ, Kang HR, Hong SU, Sung WS, Kim EJ. Efficacy and safety of electric heating moxibustion for perennial allergic rhinitis: protocol for a randomized controlled trial. Trials. 2019 Jul 19;20(1):445. doi: 10.1186/s13063-019-3550-x. PMID 31324214